CLINICAL TRIAL: NCT05618964
Title: Effects Of Deep Neck Flexor And Extensor Exercises On Pain, Range Of Motion And Muscle Strength In Mechanical Neck Pain
Brief Title: Effects Of Deep Neck Flexor And Extensor Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0154 Zahra
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Mechanical Neck Pain
Keywords: Neck muscles; Neck Pain; Muscle strength; Range of Motion
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Deep Neck Flexors & Extensors exercises (Experimental): Group A Patients will receive:
  Deep neck flexor exercises (2 set of 10 repetitions) that includes:
  * Contraction of deep neck flexor muscle in supine
  * Craniocervical flexion in supine
  Deep Neck Extensor exercises (2 set of 10 repetitions) that includes:
  * Contraction of deep neck extensors in quadruped position
  * Segmented extension movement with the head bent down onto their chest in a horizontal direction,
  Interventions: Other: Deep Neck Flexors & Extensors exercises
- Group B: Standardized Physical Therapy (No Intervention): Standardized Physiotherapy treatment will be:
  * Hot pack for 10 minutes,
  * SNAG manual therapy at Cervical spine 6 repetitions for 60 seconds.
  * Superficial neck muscles (upper trapezius, Levator scapulae, Pect.Major) stretching for 3 times with 30 seconds and
  * Neck isometrics 10 times with 6 seconds hold. Both groups will come thrice per week for a total of 4 weeks. Pre and post treatment values of both groups will be analyzed

INTERVENTIONS:
Other: Deep Neck Flexors & Extensors exercises — Deep neck flexor exercises (2 set of 10 repetitions) that includes:
  Contraction of deep neck flexor muscle in supine Craniocervical flexion in supine
  Deep Neck Extensor exercises (2 set of 10 repetitions) that includes:
  Contraction of deep neck extensors in quadruped position Segmented extension movement with the head bent down onto their chest in a horizontal direction,
  Arms: Group A: Deep Neck Flexors & Extensors exercises

SUMMARY:
Deep cervical flexor and extensor muscles show decreased strength in patients with Mechanical neck pain. Exercises involving deep cervical muscles has improved coordination and motor control. This study aim to determine the effects of deep flexor muscle exercises along with deep extensor muscle exercises on pain, range of motion and muscle strength in mechanical neck pain.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Riphah Rehabilitation Clinic Lahore and Physiotherapy outpatient department of WAPDA Teaching Hospital Lahore. Non-probability consecutive sampling will be used to collect the data. Sample size of 36 subjects with age group between 18-40 years will be taken. Data will be collected from the patients having present complaint of Mechanical Neck pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Manual Muscle Testing (MMT) for muscle strength and Universal Goniometer (GU) for Range of motion. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Both the Groups will receive Hot Pack, superficial neck muscles stretching and Neck isometrics, while Group A will receive deep neck flexor and extensor exercises, and Group B will receive conventional treatment. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 18 and 40 years of age
* Forward Head Posture
* Manual Muscle testing (MMT) grade less than 6
* Deep Flexor strength measured by pressure biofeedback unit (20 mmHg), patients who cannot hold craniocervical flexion (indicating yes) for 10 seconds

Exclusion Criteria:

* Cervical radiculopathy
* History of whiplash injury
* History of cervical and thoracic spine surgery
* Neck pain associated with vertigo
* History of spinal osteoporosis
* Vertebral Fractures
* Tumors
* Diagnosed psychological disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | follow up on 4th week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults, including those with chronic pain.
  The NPRS is a segmented numeric version in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  The NPRS takes <1 minute to complete The NPRS is a valid and reliable scale to measure pain intensity;
  * High test-retest reliability has been (r = 0.96 and 0.95, respectively)
  * For construct validity, the NPRS was shown to be highly correlated: correlations range from 0.86 to 0.95
Manual Muscle Testing (MMT) | followup on 4th week
  Muscle strength will be assessed by Manual muscle testing. Which is scored using a 0-5 points Medical Research Council muscle strength scale. MMT is the most commonly used method for documenting impairments in muscle strength in both spine and periphery with a kappa value 0.88.
Universal Goniometer (UG) | follow up on 4th week
  A goniometer is an instrument that measures the available range of motion at a joint. To measure the range of motion physical therapists most commonly use a goniometer. It is necessary that a single notation system is used in goniometry. The neutral zero method (0 to 180- degree system) is the most widely used method. The same goniometer should always be used to reduce the chances of instrumental error. The range of motion of neck including flexion and extension will be measured by using universal goniometer that has an inter-rater reliability (ICC2, 2 = 0.79 to 0.92) for cervicle region.
Pressure Biofeedback unit | follow up on 4th week
  Pressure biofeedback unit if placed under the suboccipital region and the pressure cuff is inflated to a pressure of 20 mmHg in order to fill the space of the cervical lordosis and the subject asked to perform a gentle head-nodding action of craniocervical flexion (indicating yes). Maximum pressure increase above the baseline upto 10 mmHg achieved and held for 10 seconds is defined as strength of deep cervical flexors.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Fandim JV, Nitzsche R, Michaleff ZA, Pena Costa LO, Saragiotto B. The contemporary management of neck pain in adults. Pain Manag. 2021 Jan;11(1):75-87. doi: 10.2217/pmt-2020-0046. Epub 2020 Nov 25. PMID 33234017
- [Background] Gonzalez Rueda V, Lopez de Celis C, Barra Lopez ME, Carrasco Uribarren A, Castillo Tomas S, Hidalgo Garcia C. Effectiveness of a specific manual approach to the suboccipital region in patients with chronic mechanical neck pain and rotation deficit in the upper cervical spine: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Sep 5;18(1):384. doi: 10.1186/s12891-017-1744-5. PMID 28870191
- [Background] Masaracchio M, Kirker K, States R, Hanney WJ, Liu X, Kolber M. Thoracic spine manipulation for the management of mechanical neck pain: A systematic review and meta-analysis. PLoS One. 2019 Feb 13;14(2):e0211877. doi: 10.1371/journal.pone.0211877. eCollection 2019. PMID 30759118
- [Background] Rodriguez-Sanz J, Malo-Urries M, Lucha-Lopez MO, Lopez-de-Celis C, Perez-Bellmunt A, Corral-de-Toro J, Hidalgo-Garcia C. Comparison of an exercise program with and without manual therapy for patients with chronic neck pain and upper cervical rotation restriction. Randomized controlled trial. PeerJ. 2021 Nov 24;9:e12546. doi: 10.7717/peerj.12546. eCollection 2021. PMID 34900443
- [Background] Suvarnnato T, Puntumetakul R, Uthaikhup S, Boucaut R. Effect of specific deep cervical muscle exercises on functional disability, pain intensity, craniovertebral angle, and neck-muscle strength in chronic mechanical neck pain: a randomized controlled trial. J Pain Res. 2019 Mar 7;12:915-925. doi: 10.2147/JPR.S190125. eCollection 2019. PMID 30881101
- [Background] Blomgren J, Strandell E, Jull G, Vikman I, Roijezon U. Effects of deep cervical flexor training on impaired physiological functions associated with chronic neck pain: a systematic review. BMC Musculoskelet Disord. 2018 Nov 28;19(1):415. doi: 10.1186/s12891-018-2324-z. PMID 30486819
- [Background] Alghadir AH, Iqbal ZA. Effect of Deep Cervical Flexor Muscle Training Using Pressure Biofeedback on Pain and Forward Head Posture in School Teachers with Neck Pain: An Observational Study. Biomed Res Int. 2021 May 22;2021:5588580. doi: 10.1155/2021/5588580. eCollection 2021. PMID 34095302
- [Background] Gimenez-Costa M, Schomacher J, Murillo C, Blanco-Hernandez T, Falla D, Lluch E. Specific versus non-specific exercises for the neck extensor muscles in women with chronic idiopathic neck pain: A randomized controlled trial. Musculoskelet Sci Pract. 2022 Aug;60:102561. doi: 10.1016/j.msksp.2022.102561. Epub 2022 Apr 6. PMID 35421696
- [Background] Iqbal ZA, Alghadir AH, Anwer S. Efficacy of Deep Cervical Flexor Muscle Training on Neck Pain, Functional Disability, and Muscle Endurance in School Teachers: A Clinical Trial. Biomed Res Int. 2021 Jan 13;2021:7190808. doi: 10.1155/2021/7190808. eCollection 2021. PMID 33521131
- [Background] Sikka I, Chawla C, Seth S, Alghadir AH, Khan M. Effects of Deep Cervical Flexor Training on Forward Head Posture, Neck Pain, and Functional Status in Adolescents Using Computer Regularly. Biomed Res Int. 2020 Oct 5;2020:8327565. doi: 10.1155/2020/8327565. eCollection 2020. PMID 33083487